CLINICAL TRIAL: NCT04166201
Title: Evaluation of Double Mesh Modification of Chevrel's Technique in Management of Midline Incisional Hernia
Brief Title: Double Mesh Modification of Incisional Hernia Can be Effective Without Severe Local Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hazem Nour Abdellatif, Assistant professor, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: modified chevrel technique
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Incisional Hernia of Midline of Upper Abdomen; Incisional Hernia of Midline of Lower Abdomen; Incisional Hernia of Midline of Abdomen

STUDY DESIGN:
Intervention Model Description: 22 patients with Incisional Hernia of Midline of the abdomen underwent hernioplasty by double mesh modification of Chevrel's technique follow up carried out for around 2 years for hernia recurrence pain early and late postoperative complications
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- modified chevrel technique (Other): hernioplasty done with double mesh modification of chevrels technique
  Interventions: Procedure: double mesh hernioplasty with modified chevrel's technique

INTERVENTIONS:
Procedure: double mesh hernioplasty with modified chevrel's technique — hernioplasty done by modification of the chevrel's technique , no dissection further than 1 cm of the midline laterally, the medial flaps of the anterior rectus sheath is dissected of the anterior surface of the rectus abdominis muscle and sutured together reforming the posterior rectus sheath , one polypropylene mesh was fixed over the posterior rectus sheath and the other was tailored to raw area of the rectis abdominis muscle and sutured to the lateral free edges of the anterior rectus sheath

SUMMARY:
22 patients of incisional hernia underwent treatment by double mesh modification of the original Chevrel's technique the primary outcome was recurrence, skin necrosis secondery out come was pain hematoma seroma

DETAILED DESCRIPTION:
This study is a clinical trial carried out on 22 patients with midline incisional hernia, using the double mesh modification of Chevrel's technique, all the procedures were performed by the same group of surgeons.

The exclusion criteria were American Society of Anesthesiologists (ASA) 3, and 4, inflammatory bowel disease, urgent setting, recurrences and previous abdominal neoplasms with high risk of local recurrence (rectal cancer). All patients were informed and consented before recruitment in the study All patients received an intravenous antibiotic prophylaxis with subcutaneous administration of fractionated heparin before surgery when indicated.

Surgical technique All patients were operated on with the double mesh modification of Chevrel's technique. The previous scar was excised then, dissection of the subcutaneous space was performed deep to the neck of the hernia, not wider than 1cm from the edges of the defect, then the sac was opened and resected, the defect size was measured, the skin and subcutaneous tissue was dissected off the anterior rectus sheath only allowing dissection of an anterior rectus sheath flap just sufficient to close the defect without tension After that a bilateral longitudinal incisions was done on the anterior surface of the anterior rectus sheath and a medial anterior rectus sheath flap was dissected off the rectus abdominis muscle, both recti muscles was dissected off the posterior rectus sheath opening the retrorectus space, each of the medial anterior rectus sheath flaps was sutured to that of the other side with slowly absorbed sutures closing the defect without any tension and reforming the posterior rectus sheath

A sizable prolene mesh was fixed with prolene sutures in the retrorectus space spreading between lateral ends of the space and tunneled up 4 cm in the retrorectus space far from vertical edges of the defect,Then the anterior rectus sheath was closed using a prolene mesh tailored to the size of the space between the lateral flaps of both sides and sutured to the edges of the lateral flaps with interrupted non absorbable sutures.

suction drain is left in site, subcutaneous tissue was closed with Vicryl (3\0) , skin was closed with prolene (3\0), drain was removed when the amount of drainage is below 30 ml \ day .

Data of the patients as demographic data, preoperative investigations, operative findings as defect size, operative time, early postoperative data as viability of skin flaps, wound infection, seroma and early hernia recurrence, late postoperative data as hernia recurrence. All data were collected, properly presented and analyzed using the SPSS package 22.

ELIGIBILITY:
Inclusion Criteria:

• adult with midline incisional hernia

Exclusion Criteria:

* (ASA) 3, and 4,
* inflammatory bowel disease,
* urgent setting,
* recurrences and previous abdominal neoplasms with high risk of local recurrence (rectal cancer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
recurrence of the hernia | 2 years
  the incisional hernia recurs back measured by clinical examination or abdominal CT
necrosis of the edges of the wound | 1 week
  gangrene of the medial edges of the midline incision after dissection of the skin and subcutaneous tissue off the rectus sheath measured by clinical examination

SECONDARY OUTCOMES:
seroma | 1 week
  presence of serous fluid collection in the subcutaneous space measured by superficial probe ultrasound examination
hematoma | 1 week
  blood collection around the mesh prosthesis measured by superficial probe ultrasound examination
abdominal wall pain | 1 year
  pain related to the surgical wound or the mesh prosthesis fixation sutures , measured by visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig Faculty of Medicine, Zagazig, Sharqya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided